CLINICAL TRIAL: NCT01089686
Title: Utility of Chronic Cerebrospinal Venous Insufficiency Percutaneous Angioplasty for Multiple Sclerosis: The Albany Vascular Group Study (Liberation Study)
Brief Title: Study To Evaluate Treating Chronic Cerebrospinal Venous Insufficiency (CCSVI) in Multiple Sclerosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Manish Mehta, MD (Other)
Collaborators: Center for Vascular Awareness, Albany, New York (Other)
Responsible Party: Sponsor-Investigator, Manish Mehta, MD, Principal Investigator, The Vascular Group, PLLC
Organization: The Vascular Group, PLLC (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: LS10-01
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Multiple Sclerosis
Keywords: Chronic Cerebrospinal Venous Insufficiency
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venoplasty (treatment) (Active Comparator): Patients will be randomized to treatment or non-treatment arm with a 2:1 ratio. Patients who meet the inclusion/exclusion criteria and who are randomized to the treatment arm of the study will receive venoplasty at the time of the diagnostic venogram.
  Interventions: Procedure: Venoplasty
- Sham procedure (non-treatment) (Sham Comparator): Patients will be randomized to treatment or non-treatment with a 2:1 ratio. Patients who meet the inclusion/exclusion criteria and who are randomized to the non-treatment arm of the study will receive the diagnostic venogram only.
  Interventions: Procedure: Sham procedure (non-treatment)

INTERVENTIONS:
Procedure: Venoplasty — Venous access is obtained from the groin through the femoral vein. The catheter will be advanced into the veins in the neck and chest. Angiographic images will be taken of the extracranial venous system as well as the azygous vein. These images will be used to confirm CCSVI. Venoplasty is performed by inserting an additional catheter with a balloon at the tip. The balloon will be inflated to open the vessel. Once dilation of the vessel is confirmed, the venous sheath will be removed and manual compression applied to the groin access.
  Arms: Venoplasty (treatment)
Procedure: Sham procedure (non-treatment) — Venous access is obtained from the groin through the femoral vein. The catheter will be advanced into the veins in the neck and chest. Angiographic images will be taken of the extracranial venous system as well as the azygous vein. These images will be used to confirm CCSVI. Since the patient has been randomized to the non-treatment arm of the trial, the procedure will end without venoplasty. After completion of the diagnostic venogram, the venous sheath will be removed and manual compression applied to the groin access.
  Arms: Sham procedure (non-treatment)

SUMMARY:
This is a single center, multispecialty, randomized double blind placebo control feasibility clinical trial. The purpose is to evaluate the safety, feasibility and efficacy of percutaneous transluminal angioplasty in treating extracranial venous obstructive lesions, and its influence on the clinical outcomes of Multiple Sclerosis (MS) patients that have been found to have chronic cerebrospinal venous insufficiency (CCSVI).

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old or greater and less than or equal to 65 years of age
* Score of 0 to 7 on the EDSS scale
* Diagnosis of relapsing remitting or secondary progressive Multiple Sclerosis by a neurologist and confirmed by one of the independent study neurologists
* Presence of greater than or equal to 50 percent stenosis of the extracranial veins as determined by venogram
* Informed consent signed by patient

Exclusion Criteria:

* Patient is unwilling to comply with the follow up
* Patient is pregnant
* Diagnosis of primary progressive MS by a certified neurologist confirmed by one of the study neurologists
* Presence of less than 50 percent stenosis of the extracranial veins as determined by venogram
* Presence of other medical illnesses or a psychiatric condition that in the opinion of the investigator may cause the subject to be non-compliant with the protocol requirements
* Life expectancy is less than one year
* Lack of mental capacity to consent
* Creatinine level of greater than 2.5 or is dialysis dependant
* Enrollment in another clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events | 30 days
  The evaluation of safety will be defined as the incidence of major adverse events at 30 days following the index procedure. The evaluation of feasibility and efficacy will be determined by those patients that do not have more than 50 percent restenosis within the 30 day time frame.
Neurological assessment of MS | 1 year
  An independant neurologist will assess the number of MS attacks that have occurred during one year follow up period.
MRI/MRA evaluation of MS lesions, recommended | 1 year
  Evaluation of imaging to reveal local iron content, change in MS lesions and oxygen saturation changes using conventional MRA/MRI methods by an independant radiologist.

SECONDARY OUTCOMES:
Mortality | 1 year
  All cause mortality will be evaluated through one year.
Major adverse events | 1 year
  Incidence of all major adverse events will be collected for one year.
Identification of central venous stenosis | 1 year
  Evaluation of the correlation between MRV, Duplex Ultrasound and Venogram in identifying central venous stenosis.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Mehta, MD, MPH, Principal Investigator — The Vascular Group, PLLC
Locations (1):
- The Vascular Group, PLLC, The Vascular Health Pavillion, Albany, New York, United States

REFERENCES:
- See also: The Center for Vascular Awareness — http://vaware.org